CLINICAL TRIAL: NCT01410188
Title: An Investigator-Masked, Dose-Escalation Study to Determine the Safety, Tolerability, Pharmacokinetics, and Efficacy of OPA-6566 Ophthalmic Solution in Subjects With Primary Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Safety/Efficacy Study: OPA-6566 Ophthalmic Solution in Subjects With Primary Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kubota Vision Inc. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPA-6566-101
Record Dates: First submitted 2011-07-27; First posted 2011-08-05 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-02

CONDITIONS: Primary Open-angle Glaucoma; Ocular Hypertension
Keywords: open-angle glaucoma; glaucoma; ocular hypertension; intraocular pressure
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- OPA-6566 low dose (Experimental): Treatment with OPA-6566 low dose
  Interventions: Drug: OPA-6566
- OPA-6566 medium dose (Experimental): Treatment with OPA-6566 medium dose
  Interventions: Drug: OPA-6566
- OPA-6566 high dose (Experimental): Treatment with OPA-6566 high dose
  Interventions: Drug: OPA-6566
- Latanoprost (Active Comparator): Treatment with Latanoprost
  Interventions: Drug: Latanoprost
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- OPA-6566 additional dose (Experimental): Treatment with OPA-6566 additional dose
  Interventions: Drug: OPA-6566

INTERVENTIONS:
Drug: OPA-6566 — OPA-6566, 2 dosing schedules (one drop once per day for 2 weeks and twice per day for 2 weeks)
  Arms: OPA-6566 additional dose; OPA-6566 high dose; OPA-6566 low dose; OPA-6566 medium dose
Drug: Placebo — Placebo, 2 dosing schedules (one drop once per day for 2 weeks and twice per day for 2 weeks)
  Arms: Placebo
Drug: Latanoprost — Latanoprost (one drop once per day for 4 weeks)
  Arms: Latanoprost

SUMMARY:
This is a study of the safety, tolerability, pharmacokinetics (measurement of drug levels in the blood), and intraocular pressure lowering effects of OPA-6566 ophthalmic solution in subjects with primary open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of bilateral primary open-angle glaucoma
* diagnosis of ocular hypertension as defined in the protocol

Exclusion Criteria:

* any form of glaucoma other than primary open-angle glaucoma in either eye
* other ocular conditions as defined by the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Safety: incidence of treatment emergent adverse events (TEAEs), vital signs, physical exam, ocular exams, electrocardiogram, ocular symptoms, laboratory tests on whole blood, serum and urine. | 28 days of treatment: visit 1 (screening), visit 2 (eligibility), visit 3 (randomization) visit 4 (Day 14), visit 5 (Day 28)

SECONDARY OUTCOMES:
Composite of Pharmacokinetics | 28 days: visit 3 (randomization); visit 4 (Day 14) ; visit 5 (Day 28)
Efficacy: measurement of change in intraocular pressure from baseline. | 28 days: visit 1 (screening); visit 2 (eligibility) ; visit 3 (randomization) , visit 4 (Day 14) ; visit 5 (Day 28)

CONTACTS AND LOCATIONS:
Overall Officials: John W Chandler, MD, Study Director — Kubota Vision Inc.
Locations (9):
- United States (9):
  - Artesia, California
  - Glendale, California
  - Roswell, Georgia
  - Louisville, Kentucky
  - Washington, Missouri
  - High Point, North Carolina
  - Maryville, Tennessee
  - Austin, Texas
  - San Antonio, Texas